CLINICAL TRIAL: NCT01710189
Title: Phase 4 Clinical Trial of Cervico-vaginal Immune Responses Following Three Right Deltoid or Right Thigh Intramuscular Immunisations With TicoVac (Tick Borne Encephalitis Virus [TBEV]) Vaccine in Adult Female Participants
Brief Title: Cervicovaginal Immune Responses to 3 Deltoid or Thigh Intramuscular (IM) TicoVac
Acronym: CRC306
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRC306
Record Dates: First submitted 2012-10-16; First posted 2012-10-19 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Tick-Borne Encephalitis
Keywords: Tick-Borne Encephalitis Virus
MeSH Terms: conditions — Encephalitis, Tick-Borne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TicoVac immunisation - right deltoid muscle (Experimental): IM immunisation right deltoid muscle
  Interventions: Drug: TicoVac
- TicoVac immunisation - upper anterolateral thigh (Experimental): IM: right upper anterolateral thigh
  Interventions: Drug: TicoVac

INTERVENTIONS:
Drug: TicoVac — Intramuscular immunisation to right deltoid muscle (Group 1) or right upper anterolateral thigh muscle (Group 2).

SUMMARY:
Many viral infections of global importance, including HIV, are transmitted across the mucosal surface of the genital tract. As immunity against these infections is likely to be primarily mediated by antibodies in mucosal secretions, developing techniques to increase the levels and persistence of antiviral antibody on mucosal surfaces may enhance the protection against a number of important infections. Preclinical studies have anatomically targeted vaccine antigens to sites where genital tract immunity is induced. This response is likely due to the ability of regional lymph Preclinical studies have anatomically targeted vaccine antigens to sites where genital tract immunity is induced. This response is likely due to the ability of regional lymph nodes to "pattern" the cell surface markers of responding vaccine specific lymphocytes with homing markers. In contrast, injecting a distant muscle (such as in the arm) which shares no anatomical relationship with the vagina, may not pattern cells with homing markers for the genital tract. Direct injection of inguinal lymph nodes is impractical in humans but intramuscular injection into the thigh will target antigens to the deep inguinal lymph nodes shared in common with the cervix/vagina.

This study will be a Phase IV randomised, single centre, open label, laboratory assessment blinded exploratory trial to assess mucosal immunogenicity following three targeted intramuscular immunisations with TicoVac vaccine. 20 subjects will be randomised to each of2 groups immunised in right deltoid or right anterolateral thigh.

Following an initial screening visit subjects will be immunised at 0, 1 and 6 months. There will be follow up visits 5 days after each immunisation and a final visit at 7 months. Blood samples and cervicovaginal secretions will be taken prior to each immunisation for immunological measures. In addition, blood samples will be taken at each immunisation and follow up visit for measurement of peripheral blood mononuclear cells.

The study is funded by ADITEC, which is a collaborative research programme that aims to accelerate the development of novel and powerful immunisation technologies for the next generation of human vaccines.

DETAILED DESCRIPTION:
The study will investigate whether targeting vaccine antigens to lymph nodes (internal iliac) which drain both the lower limb and the cervix/vagina alters the subsequent antibody response detected in the cervix/vagina, when compared with targeting vaccine antigens to unrelated lymph nodes such as those in the axilla that drain the right deltoid muscle of upper arm.

The right arm has been specifically selected as lymphatics in the right upper part of the body drains directly into the blood stream via the right lymphatic duct with no shared lymphatic connections to the rest of the body. In contrast lymph from the rest of the body ultimately drains into the thoracic duct (see figure below). By immunising the right arm the investigators can be sure that vaccine antigens and antigen presenting cells and activated lymphocytes will not pass through any lymph nodes in common with the cervix or vagina. In contrast by injecting the anterolateral thigh (right side selected for uniformity) the investigators can be sure that vaccine antigens will pass through the external inguinal lymph nodes which will also receive antigens and lymphocytes responding to vaginal or cervical infection or inflammation. The choice of right leg is just to standardise.

It is the investigators hypothesis therefore that as a result of antigen presentation and stimulation within a specifically "genital tract milieu" T &B lymphocytes leaving the external iliac nodes as a result of an immunisation into the thigh will be patterned in such a way as to more likely home back to the cervix and vagina due to the common drainage of the cervix, vagina and thigh (Figure 1) into the external iliac and lateral aortic lymph nodes. In contrast, cells leaving the axillary lymph nodes after immunisation of the right arm will enter the blood directly via the right lymphatic duct and so will not pass through any lymph nodes in common with the cervix and vagina.

The investigators will detect an effect of targeted immunisation in a number of ways:

1. By detecting increased levels of vaccine-specific antibodies in cervico-vaginal secretions as a result of more activated B cells (plasmablasts) homing back to the genital tract. IgG antibodies may be transudated from the blood but local mucosal IgG may also be produced. In contrast, mucosal IgA is most likely to be locally produced and may therefore be preferentially affected by targeted immunisation. However as individual levels of mucosal antibody vary widely between subjects, especially with IgA, the investigators will set primary endpoints on the basis of a fold-increase in antibody levels from baseline, rather than concentration. As mucosal IgG responses are generally more reliable and of greater magnitude the investigators have set the primary objective as vaccine-specific mucosal IgG after all three immunisations. Vaccine-specific mucosal IgA responses after all three immunisations are the secondary objective. The study has been powered on the basis of the investigators limited experience with similar vaccines to detect a doubling of proportions of responders for IgG and IgA. The investigators have based the fold-increase in vaccine-specific mucosal IgG and IgA on the investigators limited experience with a similar vaccine injected into the arm(7).

   In addition, the investigators will measure changes in other variables that are exploratory in nature as assays and quantification are less well established:
2. By detecting a "mucosal" pattern of B cell responses in the blood with increased numbers of vaccine-specific B cells after genital targeted immunisation.
3. By detecting differences in the cell surface phenotypic markers on vaccine-specific lymphocytes indicating a mucosal origin.

There will be two treatment groups:

* Group 1 will receive the vaccine in the right deltoid muscle (upper arm) which drains to unrelated lymph nodes in the axilla.
* Group 2 will receive the vaccine in the upper anterolateral right thigh, from which antigens will be expected to drain to the inguinal lymph nodes that also drain the cervix/vagina.

To ensure complete disconnection of draining lymph nodes it will always be the RIGHT arm or RIGHT leg that is immunised.

It is hypothesised that targeting the internal iliac nodes will lead to an enhanced mucosal antibody response in the cervix/vagina, which will be detected by increased vaccine-specific IgA in cervico-vaginal secretions collected in a Softcup. In addition, lymphocytes (B and T cells) from external iliac lymph nodes may carry surface markers associated with mucosal homing and secrete different combinations of cytokines (Th17) than those emanating from axillary nodes which will express a systemic phenotype. This can be detected by flow cytometry, ELISPOT after bead separation using phenotypic markers, and other immunological assays.

Immune response readouts will be IgG and IgA antibodies against the TBEV antigens in the vaccine, comparing the two groups at the time point when the peak response is expected (28 days after third immunisation).

As the investigators wish to investigate the ability of the vaccine to specifically prime subjects in a targeted way, participants must be naive to the vaccine antigens and so must not have had the vaccine or TBEV infection before. Therefore the investigators will use TicoVac - a TBEV vaccine licenced in the UK that UK adults have not generally received, as TBEV infection is not endemic in the UK. TicoVac is widely used in central and eastern Europe where TBEV is endemic but extremely uncommon, and is offered to travellers from UK to endemic areas who are likely to engage in high risk activity (hiking, trekking).

Mucosal responses against TBEV are not relevant as TBEV is transmitted by tick bites. Immune responses to TicoVac will act as a model for other vaccines in which the mucosal antibody response in the vagina is of relevance to block infection (e.g. HIV, HPV, HSV) and in which targeted immunisation may increase efficacy.

Although strictly speaking the induction of anti-TBEV antibodies in cervico-vaginal secretions is of no relevance to the efficacy of the TicoVac vaccine against a blood-injected virus, the investigators have designated them as parameters of efficacy in this model of targeted immunisation.

The purpose of this human immune physiology study is to use TBEV vaccine as a model neoantigen to investigate immune readouts after antigen targeting. The collection of adverse event or safety data is therefore not relevant to the study objectives and there will be no systematic collection of safety data, other than those required for a Risk Assessed "Type A" CTIMP (SUSAR reporting to MHRA/REC/Concerned Investigators, Annual List of Suspected Serious Adverse Reactions as part of the Annual Safety Report/Development Safety Update Report).

ELIGIBILITY:
Inclusion criteria

* Women aged between 18 and 49 years on the day of screening.
* Available for follow-up for the duration of the study.
* Willing and able to give written informed consent.
* Agree to abstain from donating blood during and for three months after the end of their participation in the trial, or longer if necessary.
* Willing to abstain from vaginal intercourse for 12 hours prior to cervico-vaginal secretions sampling.

Exclusion criteria

* Previous immunisation with a TBEV vaccine or history of TBEV infection.
* Previous immunisation with a Yellow Fever or Japanese B encephalitis vaccine, or history of infection with Yellow fever, Japanese B encephalitis, hepatitis C and dengue infection (as antibodies against these viruses cross react with TBE). Immunisation with Yellow Fever or Japanese B encephalitis vaccine or diagnosis of any of these infections during the study period will exclude the subject.
* Intention to travel to an area requiring immunisation against Japanese B encephalitis within 40 days and yellow fever within 10 days of the expected last visit(as Japanese B encephalitis vaccine requires two immunisations 28 days apart and must be completed within 10 days of departure. Yellow Fever vaccination becomes effective 10 days after a single immunisation)
* Any Intra Uterine Contraceptive Device (as this contraindicates with use of the Softcup).
* Pregnant or lactating at time of screening or immunisations.
* Known hypersensitivity to the vaccine active substance, any of the excipients, or the production residues (formaldehyde, neomycin, gentamicin, protamine sulphate).
* Latex allergy.
* Severe hypersensitivity to egg and chick proteins ("severe" means anaphylactic reaction after oral ingestion of egg protein - other reactions are not exclusions).
* Clinically relevant abnormality on history including uncontrolled infection; autoimmune disease, immunodeficiency, or pre-existing cerebral disorders.
* Any drugs and categories of drugs listed in Appendix 1, by the routes indicated, and at any time during the study period, or for the period preceding screening indicated in Appendix 1.

Any medications that are not listed in Appendix 1,or any over-the-counter treatments are not excluded.

Receipt of vaccines other than TBEV vaccines is not excluded. If other injectable vaccines are to be given during the study period, administration should preferably be into different limbs from the study vaccine.

* Receipt of blood products or immunoglobin within 3 months of screening.
* Participation in another trial of a medicinal product, completed less than 90 days prior to visit 2.
* Unable to read and speak English to a fluency level adequate for the full comprehension of procedures required in participation and consent.
* Unlikely to comply with protocol.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Primary: Proportion of subjects with a 15-fold or greater increase from pre-immunisation levels of anti-TBEV IgG in cervico-vaginal secretions at 28 days after final immunisation. | 28 weeks
  To determine whether immunisations in the anterolateral right thigh increases the proportion of subjects with a 15-fold or greater increase from pre-immunisation levels of anti-TBEV IgG in cervico-vaginal secretions at 28 days after final immunisation when compared with immunisations in the right arm

SECONDARY OUTCOMES:
Secondary: Proportion of subjects with a 2-fold or greater increase from pre-immunisation levels of anti-TBEV IgA in cervico-vaginal secretions at 28 days after final immunisation | 28 weeks
  To determine whether immunisations in the anterolateral right thigh increases the proportion of subjects with a 2-fold or greater increase from pre-immunisation levels of anti-TBEV IgA in cervico-vaginal secretions at 28 days after final immunisation when compared with immunisations in the right arm

CONTACTS AND LOCATIONS:
Overall Officials: David JM Lewis, Principal Investigator — University of Surrey
Locations (1):
- Surrey CRC, Egerton Road, Guildford, Surrey, United Kingdom

REFERENCES:
- See also: Surrey Clinical Research Centre website — https://crc.surrey.ac.uk/